CLINICAL TRIAL: NCT04755660
Title: Behavioral Intervention and Home-based Resistance Training to Increase Physical Activity and Muscle Strength in Patients With Type 2 Diabetes: A Randomized Clinical Trial
Brief Title: Home-based Resistance Training to Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Taiwan Nurses Association (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-11-004B
Record Dates: First submitted 2021-01-31; First posted 2021-02-16 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Resistance exercise; Muscle strength
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise behavior change group (EBCG) (Experimental): Behavior Change Theory-based intervention + Resistance Exercise
  Interventions: Behavioral: Exercise behavior change for resistance exercise
- Elastic band resistance exercise group( EBRG) (Active Comparator): Elastic Band Resistance Exercise
  Interventions: Behavioral: Exercise behavior change for resistance exercise
- Usual care (UC) (Sham Comparator): usual care: exercise education
  Interventions: Behavioral: Exercise behavior change for resistance exercise

INTERVENTIONS:
Behavioral: Exercise behavior change for resistance exercise — The intervention includes motivational interviews and self-efficacy theory-based exercise behavior and home-based resistance exercise intervention (by Elastic Band or non- Elastic Band ), and 3 follow-up telephone calls. The usual care group will receive exercise counseling.

SUMMARY:
The purpose of this study is to compare motivational interviews and self-efficacy theory-based exercise behavior and home-based resistance exercise (elastic band to non-elastic band) to improve physical activity, muscle strength, body composition, and self-efficacy of exercise in type 2 diabetic patients. The effectiveness of performance and exercise compliance.

DETAILED DESCRIPTION:
This study adopts an experimental research design. A total of 90 cases of type 2 diabetes who are not exercising regularly are recruited from the outpatient clinic of the Metabolism Department of a medical center in the north to participate in the study. Blocks 6, and 12 (Block) are randomly assigned. The research subjects were assigned to the behavior change and resistance exercise group, and home-based resistance exercise( with elastic band), and the control group. The behavior changes and resistance exercise group received motivational interviews and self-efficacy theory-based exercise behavior changes and resistance exercise guidance intervention, home resistance exercise. the group received home elastic band resistance exercise training, and the control group received regular exercise guidance. The three groups received data collection of physical activity, muscle strength, body composition, physical activity function, and exercise self-efficacy in the pre-test, the sixth week, and the twelfth week. During the study period, the exercise log was used to collect the mediating variable about exercise compliance (Time × frequency) data collection. This study compares the effectiveness of motivational interviews and self-efficacy theory-based exercise behavior intervention and home resistance exercise training programs. The result will show an empirical evidence for type 2 diabetic patients to increase physical activity and muscle strength in the future, and will also apply to training of muscle strengthening in diabetes and other chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 2
* age >50 years old
* sedentary lifestyle (PASE questionnaire leisure time physical activities score female <30 points, male <40 points)

Exclusion Criteria:

* severe congestive heart failure (New York Heart Association Functional Class III and IV)
* severe renal failure (estimated Glomerular Filtration Rate < 15 mL/min/1.73m2)
* stroke ((The National Institutes of Health Stroke Scale > 15)
* Peripheral Arterial Occlusive Disease
* Foot ulcer over 6 month
* Severe muscle diseases and rheumatoid arthritis
* Cognitive or mental disorders who cannot understand and cooperate with the exercise plan
* those who are accessed by the doctor to be avoided for exercise

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsae -Jyy Wang, Professor, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mori H, Kuroda A, Matsuhisa M. Clinical impact of sarcopenia and dynapenia on diabetes. Diabetol Int. 2019 Jun 19;10(3):183-187. doi: 10.1007/s13340-019-00400-1. eCollection 2019 Jul. PMID 31275784
- [Background] Nomura T, Kawae T, Kataoka H, Ikeda Y. Aging, physical activity, and diabetic complications related to loss of muscle strength in patients with type 2 diabetes. Phys Ther Res. 2018 Nov 30;21(2):33-38. doi: 10.1298/ptr.R0002. eCollection 2018. PMID 30697507
- [Background] Lee J, Kim D, Kim C. Resistance Training for Glycemic Control, Muscular Strength, and Lean Body Mass in Old Type 2 Diabetic Patients: A Meta-Analysis. Diabetes Ther. 2017 Jun;8(3):459-473. doi: 10.1007/s13300-017-0258-3. Epub 2017 Apr 5. PMID 28382531
- [Background] Mogre V, Johnson NA, Tzelepis F, Paul C. Barriers to diabetic self-care: A qualitative study of patients' and healthcare providers' perspectives. J Clin Nurs. 2019 Jun;28(11-12):2296-2308. doi: 10.1111/jocn.14835. Epub 2019 Mar 6. PMID 30791160
- [Background] Kim YH, Kim KI, Paik NJ, Kim KW, Jang HC, Lim JY. Muscle strength: A better index of low physical performance than muscle mass in older adults. Geriatr Gerontol Int. 2016 May;16(5):577-85. doi: 10.1111/ggi.12514. Epub 2015 May 28. PMID 26017097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cases were recruited at a medical center's metabolism, internal medicine outpatient clinics, and regional general clinics in Taiwan. The study received 254 referral cases, of which 9 were excluded because they did not meet the included conditions. From January 23 to December 10, 2019
Groups:
- EBCG: Exercise behavior change group (EBCG): Study subjects received one-on-one motivational interviewing-based exercise coaching and home resistance exercise training. Research subjects can choose dumbbells, kettlebells, body weights, or fitness equipment according to individual preferences, and perform resistance exercises at least 3 days a week. The total resistance exercise time every day reaches 30 minutes, including the warm-up period, exercise period, and stretching period. Starting with an intensity of 50%-60% 1RM.
- Control Group: The diabetes health teacher will provide written information and an oral explanation of diabetes exercise for about 15 minutes.
- EBRG: Elastic band resistance exercise group( EBRG): The patient receives one-to-one individual guidance on the essentials of elastic band exercise in the outpatient clinic, and the patient is asked to teach back until the patient can safely and correctly use the elastic band to perform various movements. The interventional practitioner evaluates the patient's muscle strength and provides a Thera-Band® elastic band with appropriate resistance based on the individual differences of the case. Starting with a resistance that the patient can repeat 10-12 times before feeling fatigued, the home-based elastic band resistance exercise is performed three times a week. , at least 30 minutes each time.
Period: Overall Study
Arm/Group | EBCG | Control Group | EBRG
Started | 29 | 31 | 30
Completed | 28 | 29 | 28
Not Completed | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Group: received care as usual
- EBCG: Exercise behavior change group (EBCG)
- EBRG: Elastic band resistance exercise group( EBRG)
- Total: Total of all reporting groups
Arm/Group | Control Group | EBCG | EBRG | Total
Number analyzed (Participants) | 31 | 29 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 18 | 42
  >=65 years | 20 | 16 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.61 (7.68) | 66.86 (9.53) | 62.77 (7.87) | 65.76 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 18 | 47
  Male | 16 | 15 | 12 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 31 | 29 | 30 | 90
Region of Enrollment [Number; unit: participants]
  Taiwan | 31 | 29 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity
Description: Physical activity measured leisure-time physical activity for 7 days by Physical Activity Scale for the Elderly (PASE).PASE was self-administered occupational, household, and leisure physical activities. Participants were asked about the intensity, frequency, and duration of a variety of activities, including walking; strenuous, moderate, and light sports; muscle strength and endurance; occupational activities that included standing or walking; lawn work and gardening; caring for another person; home repairs; and heavy and light housework over the previous 7 days. The frequency and duration of each activity were multiplied by an empirically derived item weight and summed to compute the total PASE score activity.15 The PASE questions work-related, household, and leisure time activities for the 7 days preceding the interview. The score is continuous, ranges from 0 to 793, and higher values indicate a more active individual.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | EBCG | EBRG
Number analyzed (Participants) | 31 | 29 | 30
score on a scale | 59.98 (52.94) | 48.21 (63.77) | 59.43 (46.10)

2. Secondary Outcome: Hand Grip Strength(kg)
Description: Hand Grip strength bilateral Grip strength will be measured using a Jamar dynamometer by asking the patient to squeeze the dynamometer handle with each hand third alternately, starting with the right hand using a standardized protocol. A brief break of approximately 1 min will be allowed between each measurement, and the maximum value will be recorded in kilograms (kg). The relative test-retest reliability of grip-strength measures obtained by dynamometry was good to excellent (intra-class correlation coefficients > 0.80) (Bohannon,2017).ICC of the test-retest with one single operator ranged from 0·60 (0·37-0·83) for the ankle extensors to 0·85 (0·74-0·95) for the elbow flexors.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Kg
Groups:
- Control Group: received care as usual usual care: exercise education
  Exercise behavior change for resistance exercise: The intervention includes motivational interviews and self-efficacy theory-based exercise behavior and home-based resistance exercise intervention (by Elastic Band or non- Elastic Band ), and 3 follow-up telephone calls. The usual care group will receive exercise counseling.
- EBCG: Exercise behavior change group(EBCG) Behavior Change Theory-based intervention + Resistance Exercise
  Exercise behavior change for resistance exercise: The intervention includes motivational interviews and self-efficacy theory-based exercise behavior and home-based resistance exercise intervention (by Elastic Band or non- Elastic Band ), and 3 follow-up telephone calls. The usual care group will receive exercise counseling.
- EBRG: Elastic band resistance exercise group(EBRG)
Arm/Group | Control Group | EBCG | EBRG
Number analyzed (Participants) | 31 | 30 | 29
Kg | 28 (7.93) | 29.36 (10.03) | 28.22 (7.61)

3. Secondary Outcome: Body Composition
Description: In this study, body composition used bioelectrical impedance analysis (BIA) to analyze body muscle and fat data.was measured by OM-ROM HF-701 for body weight, and a body fat machine was used to measure the participants' body weight, body fat, and limb skeletal muscle ratio. The skeletal muscle rate of the whole body, arms, trunk, and feet was measured using a single frequency on four poles (a 50 kHz single frequency, measured by four guide hands and feet). The value range is 5.0~50.0%, with 0.1% as the unit. The measurements obtained from the device indicate the ratio of total skeletal muscle mass and body fat relative to body weight. The skeletal muscle weight cut-off points for sarcopenia are <37.5% for men and <32.6% for women; the cut-off points for fat rate and obesity are >29% for men and >40% for women.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Control Group | EBCG | EBRG
Number analyzed (Participants) | 31 | 29 | 30
percentage of body weight
  skeletal muscle ratio | 25.02 (3.74) | 23.87 (3.7) | 24.74 (3.51)
  body fat ratio | 27.88 (7.25) | 27.09 (7.45) | 27.07 (7.06)

4. Secondary Outcome: Self-efficacy
Description: self-efficacy about exercise will measured by Chinese version of the self-efficacy for exercise (SEE-C) scale . It was designed to test people's confidence to continue exercising in the face of barriers to exercise.The participants will instruct to listen to the statement and then choose an option from 0 (not confident) to 10 (very confident). The scale was scored by summing the numerical ratings for each response and dividing the total by the number of non-missing responses. The mean scores for the self-efficacy of exercise ranged from 0 to 10, with the higher scores representing greater exercise self-efficacy.SEE-C has acceptable levels of reliability and validity for the scale when used with older people in Taiwan.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | EBCG | EBRG
Number analyzed (Participants) | 31 | 29 | 30
score on a scale | 2.53 (2.96) | 4.0 (2.49) | 3.72 (2.68)

5. Secondary Outcome: Physical Performance_30-s Chair Stand Test.
Description: Physical performance was a 30-s chair stand test.
  30-s chair stand test: Participants were instructed to rise as quickly as possible from a seated position, with full body weight on the chair, to a standing posture, with their legs fully extended while keeping their arms folded across their chest. The 30CST measures the maximal number of chair stands completed during 30 seconds of the test.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: chair stands
Arm/Group | Control Group | EBCG | EBRG
Number analyzed (Participants) | 31 | 29 | 30
chair stands | 12.35 (3.96) | 13.76 (3.91) | 13.97 (4.13)

6. Secondary Outcome: Hemoglobin A1c
Description: Glycosylated Hemoglobin was taken some days(around 1 week) before the clinical visit. HbA1c was measured by a commercial pathology laboratory using standard assays.
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total haemoglobin
Arm/Group | Control Group | EBCG | EBRG
Number analyzed (Participants) | 31 | 29 | 30
percentage of total haemoglobin | 7.24 (1.03) | 7.16 (0.89) | 7.11 (0.85)

7. Secondary Outcome: Physical Performance _6-meter Walking Speed.
Description: 6-meter walking speed: Participants walked twice at their usual pace over a 6-meter course. Time in seconds was recorded between the 2nd and the 4th meter. Distance (m) divided by time (s) was used to calculate walking speed. Slow gait speed was defined using AWGS 2019 reference value of < 1.0 m/s
Time Frame: Change from Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: meter/second
Arm/Group | Exercise Behavior Change Group (EBCG) | Elastic Band Resistance Exercise Group( EBRG) | Usual Care (UC)
Number analyzed (Participants) | 29 | 30 | 31
meter/second | 0.09 (0.18) | 0.18 (0.64) | 0.13 (0.22)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Group | EBCG | EBRG
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT04755660/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT04755660/SAP_001.pdf